CLINICAL TRIAL: NCT03331081
Title: Effects of Bladder Training and Pelvic Floor Muscle Training on the Symptomatology of Overactive Bladder Syndrome - a Randomized Controlled Clinical Trial
Brief Title: Effects of Bladder Training and Pelvic Floor Muscle Training on the Symptomatology of Overactive Bladder Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Letícia de Azevedo Ferreira, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder Syndrome
MeSH Terms: interventions — 4,4',5'-trimethylazapsoralen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Bladder Training (Experimental): Patients will receive verbal instructions on bladder function (filling and bladder emptying phases), pelvic floor musculature on bladder function; orientation on urinary positioning and habits (urinary frequency); and the definition and major risk factors responsible for urinary incontinence.
  Interventions: Other: Bladder Training
- Group TMAP (Active Comparator): In this group the patients will perform TMAP in isolation. The training protocol aims at the work of strength and muscular hypertrophy, with concentric-isometric muscular action and load of 100% of the maximum voluntary contraction.
  Interventions: Other: TMAP
- Group Bladder Training + TMAP (Active Comparator): In this group, the patients should perform the proposed exercises for the Bladder Training Group and the exercises proposed for the TMAP Group. The training protocol of this group will consist of exercises that have as objectives: to improve the control over the urgency and urge-incontinence; increase bladder capacity, and thus prolong the intervals between urinations; to restore confidence in bladder control; and improve MAP strength and hypertrophy.
  Interventions: Other: Bladder Training + TMAP

INTERVENTIONS:
Other: Bladder Training — The patient will participate in a class in which the physiotherapist will provide the following information: on the anatomy and function of the MAP, using figures; on bladder function; guidelines on the positioning and voiding habits and the definition and main risk factors responsible for urinary incontinence. The bladder training will consist of a program of time micturition to increase bladder capacity and the interval between urinations. Urge suppression strategies will be targeted, and include distraction, relaxation, breathing, and MAP contraction (quick flicks).
  Arms: Group Bladder Training
Other: TMAP — There will be 36 monthly series of home training (totaling at the end of the 3 months of treatment 108 series) performed 3x / week, 3x / day. The training protocol consists of three daily TMAP series. One series consists of 8 maximum voluntary contractions, with maintenance of the contraction of 6 to 10 seconds (type I muscle fibers), with twice the rest time between contractions, followed by three to five rapid contractions (muscle fibers type II ). The protocol will total 24 contractions of MAP per day performed, which will be divided in the morning (8 contractions), late (8 contractions) and night (8 contractions).
  Arms: Group TMAP
Other: Bladder Training + TMAP — Will perform the exercises of the bladder training group and the TMAP in an associated way.
  Arms: Group Bladder Training + TMAP

SUMMARY:
The question is whether vesical training and TMAP can be used in isolation without treatment of overactive bladder syndrome? ALSO will be evaluated in urinary symptoms, a function of the MAP, a quality of life and a satisfaction of the women with the treatment offered.

DETAILED DESCRIPTION:
Bladder training includes as resources the educational program, lifestyle modifications, as a strategy to suppress urgency and as programmed urges to improve the control of urgency and incontinence; increase bladder capacity, and thus prolong the intervals between such as urination; giving the patient a confidence in the bladder control. Already, a justification for the use of TMAP is a contraction of the pelvic floor muscles (MAP) inhibits detrusor contraction, improving the symptoms of detrusor overactivity.

ELIGIBILITY:
Inclusion Criteria:

* Women with IUU and / or IUM with a predominance of urinary urgency, capable of contracting MAPs adequately, and who agree to participate in the study, signing the Informed Consent Form.

Exclusion Criteria:

* Women with a diagnosis of glaucoma, myasthenia gravis, urinary tract obstruction, neurological and chronic-degenerative diseases, decompensated diabetic patients and patients with complete denervation of the pelvic floor, pregnancy, abnormal genital bleeding, impairment of cognition, inability to fill in the diary voiding, genital dystopias beyond the vaginal introitus and urethral sphincter defect. Patients may not be in use or have used anticholinergics, tricyclic antidepressants or local hormone therapy within the six months prior to the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-11-25 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of subjective cure | At the end of 3 months of supervised treatment
  We consider it "satisfied" when the patient does not want another treatment, and "dissatisfied" when the patient wants another treatment option.

SECONDARY OUTCOMES:
BMI | At the initial evaluation of the patient before starting the 3 months of treatment
  Weight and height will be combined to report BMI in kg / m2
Urinary symptoms | At the initial evaluation of the patient before starting the 3 months of treatment
  Duration of urinary symptoms
Pregnancies and deliveries | At the initial evaluation of the patient before starting the 3 months of treatment
  Number of pregnancies and vaginal deliveries
Pad test | At the initial evaluation of the patient before starting the 3 months of treatment and the end of 3 months of supervised treatment
  The patient will be instructed to empty the bladder and place a preweighed absorbent. Afterwards, the patient will be asked to ingest 500 ml of sodium free (water) liquid during the first 15 minutes of the examination. After the rest period of 1 hour, the patient will be guided to walk for 30 minutes, in which she must climb and descend five flights of stairs for ten consecutive times. Next, a sequence of exercises will be performed: coughing vigorously for 10 times, squatting 10 times, jumping in place 10 times, and washing hands in running water for 1 minute. Once the activities are over, the absorbent will be weighed again to check for urinary loss.
V8 questionnaire | At the initial evaluation of the patient before starting the 3 months of treatment and the end of 3 months of supervised treatment
  This scale includes eight issues of urgency, incontinence, nocturia, and voiding frequency. The score for each response varies from 0 (no nuisance) to 5 (extremely uncomfortable), reaching a total of 40 points, being considered positive for SBH when the sum of the questions is equal to or greater than eight.
Voiding diary | At the initial evaluation of the patient before starting the 3 months of treatment and the end of 3 months of supervised treatment
  Patients should document how many times they go to the restroom during the day and at night, as well as the loss of urine in stressful situations (coughing, sneezing, laughter, squatting, weightlifting, walking, running), changing liner or absorbent and episodes of urgency and urgency-incontinence. The journal shall be held for a consecutive period of 24 hours, for a minimum of three consecutive days.
Quality of life | At the initial evaluation of the patient before starting the 3 months of treatment and the end of 3 months of supervised treatment
  Incontinence Quality of Life Questionnaire - I-QoL: It is composed of 22 questions organized in three domains. Limitation of human behavior; psychosocial impact; embarrassment and social embarrassment. The values added should vary between 0 and 100 points, and the lower the number obtained the greater the impact of urinary incontinence on quality of life.
MAP function | At the initial evaluation of the patient before starting the 3 months of treatment and the end of 3 months of supervised treatment
  NEW PERFECT: The examiner's fingers will be positioned approximately four centimeters from the vaginal introitus, and muscle function will be assessed. The examiner's fingers will be positioned approximately four centimeters from the vaginal introitus, and muscle function will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Letícia Ferreira, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598